CLINICAL TRIAL: NCT05181033
Title: A Phase II Randomized Trial of Lenvatinib Combined With Letrozole Versus Fulvestrant in Metastatic Estrogen Receptor (ER) Positive, HER2 Negative Breast Cancer, Who Have Progressed on First-line Aromatase Inhibitor + a CDK4/6 Inhibitor.
Brief Title: Lenvatinib+Letrozole Versus Fulvestrant in Metastatic ER+/HER2- Breast Cancer, Post Progression on Al + CDK4/6 Inhibitor
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National University Hospital, Singapore (Other)
Collaborators: Eisai Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BR01/02/21
Record Dates: First submitted 2021-11-30; First posted 2022-01-06 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Breast Cancer
Keywords: Metastatic Estrogen Receptor (ER) positive; HER2 negative; breast cancer; first-line aromatase inhibitor; CDK4/6 inhibitor
MeSH Terms: conditions — Breast Neoplasms | interventions — lenvatinib; Letrozole; Fulvestrant

STUDY DESIGN:
Intervention Model Description: This is a multi-centre study comprising two phases: a lead-in phase II (Part A) followed by a randomized phase II portion (Part B).
  Part A: Lead in phase II study A total of up to 10 patients will be enrolled. Patients will be treated with letrozole 2.5mg daily plus lenvatinib 14mg daily until disease progression or unacceptable toxicity. ' Part B: Randomised phase II study
  Patients will be randomized in a 1:1 fashion to one of 2 arms:
  * Control arm: intramuscular (IM) fulvestrant 500mg on day 1 and day 15 during cycle 1, then day 1 only from cycle 2 onwards of every 4-weekly cycle
  * Experimental arm: oral (PO) letrozole 2.5mg daily plus lenvatinib 14mg daily A total of 110 patients with ER positive breast cancer and measurable primary tumor will be enrolled over a period of 24-30 months.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control arm (Active Comparator): intramuscular (IM) fulvestrant 500mg on day 1 and day 15 during cycle 1, then day 1 only from cycle 2 onwards of every 4-weekly cycle
  Interventions: Drug: Fulvestrant
- Experimental arm (Experimental): oral (PO) letrozole 2.5mg daily plus lenvatinib 14mg daily
  Interventions: Drug: Lenvatinib + Letrozole

INTERVENTIONS:
Drug: Lenvatinib + Letrozole — Patient will receive letrozole 2.5mg daily plus lenvatinib 14mg daily until disease progression/unacceptable toxicity.
  Patient review, safety evaluations, thyroid function monitoring and urine dipstick will be done. Toxicities will be graded using NCI CTCAE toxicity grading vs 4.0. Patient should be discontinued if drug cannot be resumed within 28 days due to toxicities.
  Drugs should be withheld when subject has imminent risk to develop hypertensive crisis/has significant risk factors for severe complications of uncontrolled hypertension. Drugs can be resumed once patient received same hypertensive medications for at least 48 hours and the BP is controlled.
  Lenvatinib should be withheld for at least 1 week prior to elective surgery, at least 2 weeks after major surgery, until adequate wound healing.
  For risk of ONJ, oral dental examination and preventive dentistry should be considered prior to lenvatinib intake.
  There is no dose modifications for letrozole.
  Other Names: Lenvima
  Arms: Experimental arm
Drug: Fulvestrant — Patients will be treated with Fulvestrant 500mg injections that are administered into the muscles (intramuscularly). This is injected at 2-weekly interval for the first 3 doses, followed by 4-weekly interval dosing.
  Other Names: Faslodex
  Arms: Control arm

SUMMARY:
Based on the results of the phase Ib/II study, the investigators hypothesize that combining a RET inhibitor lenvatinib with endocrine therapy letrozole improves objective response and progression-free survival compared to fulvestrant alone in the second line setting in patients who have progressed on first line endocrine therapy incorporating a CDK4/6 inhibitor.

Letrozole and fulvestrant are anti-hormonal drugs that have been proven to have activity and are considered standard therapies for hormone receptor positive breast cancer. The purpose of this study is to determine if the combination therapy of letrozole (an anti-hormonal drug) and lenvatinib (a targeted therapy), when compared to another anti-hormonal drug fulvestrant, is effective in patients with hormone receptor positive breast cancer.

Preliminary studies have shown that approximately 50-60% of hormone receptor positive breast cancers over-express RET, and may therefore respond to treatment by a drug that blocks the RET pathway. An earlier study conducted at the National University Cancer Institute, Singapore (NCIS) on the combination of letrozole and Lenvatinib has shown promising results. Among patients in whom hormonal therapy and a CDK4/6 inhibitor no longer worked, about one-quarter of patients had meaningful disease control. The study also showed that patients tolerated the combination of Lenvatinib and letrozole well with manageable side effects.

Based on the promising findings from the earlier study, this study seeks to compare the effectiveness of lenvatinib plus letrozole with another standard anti-hormone treatment drug called fulvestrant.

In addition, investigators are studying how body reacts to the treatment as well as studying gene and protein changes in the tumour in response to treatment, which may in the future, help us tailor drug treatment for individual patients according to the patient's and/or the tumour's genetic or protein make-up.

DETAILED DESCRIPTION:
Breast cancer is the commonest cancer among females in Singapore and worldwide. Approximately 60-70% of breast cancers are hormone receptor positive and thus potentially sensitive to endocrine therapy. However, both primary and acquired resistance to endocrine therapy exists, and better combinations are constantly being explored to delay endocrine resistance and improve treatment outcome. Several known mechanisms of endocrine resistance have been proposed, and include deregulation of various components of the ER pathway itself, alterations in cell cycle and cell survival signaling molecules, and the activation of escape pathways that can provide tumors with alternative proliferative and survival stimuli.

Endocrine blockade in breast cancer can be achieved by reducing the levels of estrogens through ovarian ablation (medical, surgical, or through radiation) in pre-menopausal women or with the administration of aromatase inhibitors (AI) in post-menopausal women. Direct inhibition of estrogen receptors can be achieved by administering selective estrogen receptor modulators, such as tamoxifen, or a pure estrogen receptor antagonist such as fulvestrant. Sequential single agent endocrine therapy used to be the standard of care in advanced hormone receptor positive, HER2 negative breast cancer patients without visceral crisis and low tumor burden. However, the development of CDK4/6 inhibitors (palbociclib, ribociclib and abemaciclib) since 2014 has resulted in endocrine therapy + CDK4/6 inhibitor becoming a new standard of care in the first- or second-line setting for these patients, even in those with visceral disease (though not visceral crisis) and substantial tumor burden. The addition of CDK4/6 inhibitors has resulted in consistent improvement in progression-free survival 2-4, and a recent meta-analyses has also confirmed improvement in overall survival outcomes.

There is limited literature on the median progression-free survival (PFS) of single agent fulvestrant in patients who have failed first-line AI + CDK4/6 inhibitors. However, in several contemporary phase II/III randomized trials of second-line endocrine therapy in patients who failed prior AI (majority or all had no prior CDK4/6 inhibitors), e.g., FAKTION, SANDIPIPER, BELLE2 trials, median PFS in the control arm of single agent fulvestrant is fairly consistent at 4.5 to 5.6 months. Median PFS of fulvestrant post-progression from first-line AI + CDK4/6 inhibitors is expected to be shorter than 4.5 to 5.6 months as these patients are likely to be more endocrine-resistant. In a subgroup analysis of patients who failed prior CDK4/6 inhibitors (n=20) and who received single agent fulvestrant as second-line endocrine therapy in the phase III randomized SOLAR-1 trial, median PFS was 1.8 months and 1-year PFS was <10%.

RET is an estrogen response gene, and preclinical studies have demonstrated cross talk between RET and ER. Significant interactions between RET and ERa pathways have been described, with increased response to estrogen stimulation observed in the presence of functional RET. RET is associated with resistance to tamoxifen and aromatase inhibitors, and increased RET expression has been demonstrated in hormone resistant cell lines and primary tumors. Combined anti-estrogen and anti-RET therapy in luminal breast cancer had a greater effect on cell growth than either therapy alone. The two classes of drugs have different mechanisms of action; a RET tyrosine kinase inhibitor (TKI) reduced growth through induction of apoptosis, while anti-ERa reduced cell proliferation, forming the biologic basis for dual treatment. Dual therapy with tamoxifen and vandetinib, a RET inhibitor, resulted in greater reduction in tumor growth rate in MCF7 xenografts in mice. RET has been reported to be over-expressed in up to 75% of ER+ breast cancers (n=20), compared to only 10% of ER-negative breast cancers (n=10) in a small study.

Preclinical experiments from laboratory showed lenvatinib to have activity in ER positive breast cancer cell lines, regardless of levels of RET expression. Lenvatinib was at least additive with tamoxifen in all 6 ER positive breast cancer cell lines tested, with the combination resulting in =50% cell kill compared to single agent tamoxifen in BT474, CAMA1, and T47D cell lines supporting the potential role of lenvatinib in combination with endocrine therapy in the treatment of ER positive breast cancers.

A phase Ib with dose expansion study was carried out at the National University Cancer Institute, Singapore with the use of lenvatinib together with letrozole in the treatment of patients with estrogen receptor positive, HER2 negative breast cancer. This study was initiated in patients for neoadjuvant therapy, but expanded to include patients with metastatic breast cancer. In total, 47 patients were enrolled, among whom the first 4 patients received neoadjuvant therapy for locally advanced disease, and the remaining 43 patients received treatment in the metastatic setting. Recommended phase 2 dose of lenvatinib was established at 14mg daily in combination with letrozole 2.5mg daily. Thirty-one patients were enrolled in the dose expansion cohort at recommended phase 2 dose (RP2D).

At interim analyses, patients enrolled had a median of 4 prior lines of therapy (range 0-11), with 78.9% of patients having prior exposure to CDK4/6 inhibitor therapy. In the intention-to-treat population, an overall response rate (ORR) of 36.8% was observed, with 28.9% patients remaining progression-free (PPF) at 1 year. Among patients with partial response or stable disease, median duration of response was 16.1 months (range 5.4 to 21.7 months). Amongst these patients, 78.9% (n=30) had prior CDK4/6 inhibitor treatment, and 12 patients received CDK4/6 inhibitors as immediate prior line of therapy. In the subset of patients with prior CDK4/6 inhibitor exposure, similar encouraging results were observed, with a ORR of 26.7, 23.3% PPF at 1 year, and duration of response of 13.2 months (range 3.8 to 21.3 months).

Additionally, on-target effect, downregulation of RET expression among tumors were found to have positive RET expression at baseline. Main toxicities observed included hypertension (all grade 59%, grade3 8%), hypothyroidism (all grade 46%, grade 3 0%), and fatigue (all grade 43%, grade 3 5%), all of which were well controlled with optimal medical therapy. No grade 4-5 toxicities were observed. The promising results from the phase Ib study forms the basis of this randomized phase II study.

ELIGIBILITY:
Inclusion Criteria:

Patients may be included in the study only if patient meet all of the following criteria:

* Female, age =>18 years.
* Histologic or cytologic diagnosis of breast carcinoma.
* Estrogen receptor positive (defined as =>1% on immunohistochemical staining)
* Progressed on first-line palliative endocrine therapy plus CDK4/6 inhibitor as immediate prior line of endocrine therapy. Prior palliative letrozole is allowed.
* Only one prior line of endocrine therapy in the metastatic setting.
* No more than 1 prior line of chemotherapy in the metastatic setting.
* Measurable disease by RECIST criteria.
* ECOG 0-1.
* Estimated life expectancy of at least 12 weeks.
* Adequate organ function including the following:

  - Bone marrow: Absolute neutrophil (segmented and bands) count (ANC) =>1.5 x 109/L Platelets =>100 x 109/L

  - Hepatic: Bilirubin <= 1.5 x upper limit of normal (ULN), ALT or AST<= 2.5x ULN, (or <=5 X with liver metastases)

  - Renal: Creatinine <= 1.5x ULN
* Normal thyroid function on thyroid screen (fT4 and TSH). Patients who have thyroid dysfunction are eligible if thyroid function is optimally controlled.
* Post-menopausal women. Post-menopausal status is defined either by Age => 60 years and one year or more of amenorrhea Age <= 60 years and one year or more of amenorrhea (in the absence of ovarian suppression) and with estradiol and FSH levels consistent with menopause, Pre-menopausal women who are treated with medical ovarian suppression with post-menopausal levels of estradiol (institutional limits) at time of study entry and who will continue to be suppressed with 4-weekly LHRH agonist during study treatment may be enrolled. If these patients were previously on 12-weekly long-acting LHRH agonist, this has to be switched to 4-weekly LHRH agonist while the patient is on study treatment.
* Signed informed consent from patient or legal representative.

Exclusion Criteria:

Patients will be excluded from the study for any of the following reasons:

* HER2 positive tumors.
* Treatment within the last 30 days with any investigational drug.
* Prior therapy with fulvestrant.
* Concurrent administration of any other tumor therapy, including cytotoxic chemotherapy, hormonal therapy, and immunotherapy.
* Major surgery within 28 days of study drug administration.
* Active infection that in the opinion of the investigator would compromise the patient's ability to tolerate therapy.
* Pregnancy.
* Breast feeding.
* Serious concomitant disorders that would compromise the safety of the patient or compromise the patient's ability to complete the study, at the discretion of the investigator.
* Non-healing wound.
* Poorly controlled diabetes mellitus.
* Second primary malignancy that is clinically detectable at the time of consideration for study enrollment.
* Uncontrolled or symptomatic brain metastases, and/or brain metastases requiring steroids
* History of significant neurological or mental disorder, including seizures or dementia.
* Uncontrolled blood pressure (defined as persistent systolic BP >140 mmHg or diastolic BP>90mmHg) in spite of optimized regimen of antihypertensive medication
* Presence of proteinuria defined as 24h urine collection of grade 2 and above (protein >1.0g/24h)
* Significant cardiovascular impairment: history of congestive heart failure greater that New York Heart Association (NYHA) Class II, unstable angina, myocardial infarction or stroke within 6 months of first dose of study drug, or cardiac arrhythmia requiring medical treatment at screening.
* Bleeding or thrombotic disorders or gastrointestinal bleeding event or active hemoptysis or use of anticoagulants such as warfarin or similar agents requiring therapeutic INR monitoring, or subjects at risk of severe hemorrhage. The degree of tumor invasion/infiltration of major blood vessels should be considered because of the potential risk of severe hemorrhage associated with tumor shrinkage / necrosis following Lenvatinib therapy.
* Patients with baseline QTc interval >480ms that persists despite correction of electrolyte abnormalities and/or discontinuation of concomitant medications that are known to prolong QTc interval.

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Breast cancer study - 99.9% breast cancer patients are female. Male breast cancer is extremely rare and investigators do not intend to include this rare population
Enrollment: 120 (Estimated)
Dates: Start 2021-12-27 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) of patients treated on lenvatinib and letrozole compared to single agent fulvestrant | 30 months
  The PFS will be described using the Kaplan-Meier method and compared via logrank test.
  A total of 10 patients will be enrolled in the lead in portion of the study. If median PFS of the 10 patients is ≥4.5 months (upper limit of the 95% CI of median PFS to single agent fulvestrant in the retrospective study from NCIS), investigators will proceed to phase II randomized trial. If median PFS of the 10 patients is <3 months, study will not proceed to phase II randomized portion. If the median PFS of the 10 patients is between >3 months and <4.5 months, the study scientific committee will review and decide whether to proceed to the next part of trial. Interim analysis will be performed after 6 patients have been enrolled and the patient has been on study treatment for ≥6 months. If the PFS of all 6 patients is ≥4.5 months, investigators will move into the phase II randomized portion without the need to complete recruitment of all 10 patients into the lead-in phase II portion.

SECONDARY OUTCOMES:
Overall objective response rate (ORR) measured by RECIST 1.1 criteria of patients treated with lenvatinib and letrozole compared to single agent fulvestrant | 30 months
  The ORR rates will be compared using the exact binomial test add quantified in terms of difference in proportion as well as relative risk estimate and the associated 95% confidence intervals.
Clinical benefit rate (CBR) measured by RECIST 1.1 criteria of patients treated with lenvatinib and letrozole compared to single agent fulvestrant | 30 months
  The CBR rates will be compared using the exact binomial test add quantified in terms of difference in proportion as well as relative risk estimate and the associated 95% confidence intervals.
Overall survival (OS) of patients treated with lenvatinib and letrozole compared to single agent fulvestrant | 30 months
  The OS curves will be described using the Kaplan-Meier method and compared via logrank test.

CONTACTS AND LOCATIONS:
Overall Officials: Soo Chin Lee, Principal Investigator — National University Hospital, Singapore
Locations (1):
- Nationa University Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Osborne CK, Schiff R. Mechanisms of endocrine resistance in breast cancer. Annu Rev Med. 2011;62:233-47. doi: 10.1146/annurev-med-070909-182917. PMID 20887199
- [Background] Finn RS, Martin M, Rugo HS, Jones S, Im SA, Gelmon K, Harbeck N, Lipatov ON, Walshe JM, Moulder S, Gauthier E, Lu DR, Randolph S, Dieras V, Slamon DJ. Palbociclib and Letrozole in Advanced Breast Cancer. N Engl J Med. 2016 Nov 17;375(20):1925-1936. doi: 10.1056/NEJMoa1607303. PMID 27959613
- [Background] Tripathy D, Im SA, Colleoni M, Franke F, Bardia A, Harbeck N, Hurvitz SA, Chow L, Sohn J, Lee KS, Campos-Gomez S, Villanueva Vazquez R, Jung KH, Babu KG, Wheatley-Price P, De Laurentiis M, Im YH, Kuemmel S, El-Saghir N, Liu MC, Carlson G, Hughes G, Diaz-Padilla I, Germa C, Hirawat S, Lu YS. Ribociclib plus endocrine therapy for premenopausal women with hormone-receptor-positive, advanced breast cancer (MONALEESA-7): a randomised phase 3 trial. Lancet Oncol. 2018 Jul;19(7):904-915. doi: 10.1016/S1470-2045(18)30292-4. Epub 2018 May 24. PMID 29804902
- [Background] Goetz MP, Toi M, Campone M, Sohn J, Paluch-Shimon S, Huober J, Park IH, Tredan O, Chen SC, Manso L, Freedman OC, Garnica Jaliffe G, Forrester T, Frenzel M, Barriga S, Smith IC, Bourayou N, Di Leo A. MONARCH 3: Abemaciclib As Initial Therapy for Advanced Breast Cancer. J Clin Oncol. 2017 Nov 10;35(32):3638-3646. doi: 10.1200/JCO.2017.75.6155. Epub 2017 Oct 2. PMID 28968163
- [Background] Li J, Huo X, Zhao F, Ren D, Ahmad R, Yuan X, Du F, Zhao J. Association of Cyclin-Dependent Kinases 4 and 6 Inhibitors With Survival in Patients With Hormone Receptor-Positive Metastatic Breast Cancer: A Systematic Review and Meta-analysis. JAMA Netw Open. 2020 Oct 1;3(10):e2020312. doi: 10.1001/jamanetworkopen.2020.20312. PMID 33048129
- [Background] Jones RH, Casbard A, Carucci M, Cox C, Butler R, Alchami F, Madden TA, Bale C, Bezecny P, Joffe J, Moon S, Twelves C, Venkitaraman R, Waters S, Foxley A, Howell SJ. Fulvestrant plus capivasertib versus placebo after relapse or progression on an aromatase inhibitor in metastatic, oestrogen receptor-positive breast cancer (FAKTION): a multicentre, randomised, controlled, phase 2 trial. Lancet Oncol. 2020 Mar;21(3):345-357. doi: 10.1016/S1470-2045(19)30817-4. Epub 2020 Feb 5. PMID 32035020
- [Background] Dent S, Cortes J, Im YH, Dieras V, Harbeck N, Krop IE, Wilson TR, Cui N, Schimmoller F, Hsu JY, He J, De Laurentiis M, Sousa S, Drullinsky P, Jacot W. Phase III randomized study of taselisib or placebo with fulvestrant in estrogen receptor-positive, PIK3CA-mutant, HER2-negative, advanced breast cancer: the SANDPIPER trial. Ann Oncol. 2021 Feb;32(2):197-207. doi: 10.1016/j.annonc.2020.10.596. Epub 2020 Nov 10. PMID 33186740
- [Background] Baselga J, Im SA, Iwata H, Cortes J, De Laurentiis M, Jiang Z, Arteaga CL, Jonat W, Clemons M, Ito Y, Awada A, Chia S, Jagiello-Gruszfeld A, Pistilli B, Tseng LM, Hurvitz S, Masuda N, Takahashi M, Vuylsteke P, Hachemi S, Dharan B, Di Tomaso E, Urban P, Massacesi C, Campone M. Buparlisib plus fulvestrant versus placebo plus fulvestrant in postmenopausal, hormone receptor-positive, HER2-negative, advanced breast cancer (BELLE-2): a randomised, double-blind, placebo-controlled, phase 3 trial. Lancet Oncol. 2017 Jul;18(7):904-916. doi: 10.1016/S1470-2045(17)30376-5. Epub 2017 May 30. PMID 28576675
- [Background] Andre F, Ciruelos E, Rubovszky G, Campone M, Loibl S, Rugo HS, Iwata H, Conte P, Mayer IA, Kaufman B, Yamashita T, Lu YS, Inoue K, Takahashi M, Papai Z, Longin AS, Mills D, Wilke C, Hirawat S, Juric D; SOLAR-1 Study Group. Alpelisib for PIK3CA-Mutated, Hormone Receptor-Positive Advanced Breast Cancer. N Engl J Med. 2019 May 16;380(20):1929-1940. doi: 10.1056/NEJMoa1813904. PMID 31091374
- [Background] Boulay A, Breuleux M, Stephan C, Fux C, Brisken C, Fiche M, Wartmann M, Stumm M, Lane HA, Hynes NE. The Ret receptor tyrosine kinase pathway functionally interacts with the ERalpha pathway in breast cancer. Cancer Res. 2008 May 15;68(10):3743-51. doi: 10.1158/0008-5472.CAN-07-5100. PMID 18483257
- [Background] Plaza-Menacho I, Morandi A, Robertson D, Pancholi S, Drury S, Dowsett M, Martin LA, Isacke CM. Targeting the receptor tyrosine kinase RET sensitizes breast cancer cells to tamoxifen treatment and reveals a role for RET in endocrine resistance. Oncogene. 2010 Aug 19;29(33):4648-57. doi: 10.1038/onc.2010.209. Epub 2010 Jun 7. PMID 20531297
- [Background] Morandi A, Martin LA, Gao Q, Pancholi S, Mackay A, Robertson D, Zvelebil M, Dowsett M, Plaza-Menacho I, Isacke CM. GDNF-RET signaling in ER-positive breast cancers is a key determinant of response and resistance to aromatase inhibitors. Cancer Res. 2013 Jun 15;73(12):3783-95. doi: 10.1158/0008-5472.CAN-12-4265. Epub 2013 May 6. PMID 23650283
- [Background] Spanheimer PM, Cyr AR, Gillum MP, Woodfield GW, Askeland RW, Weigel RJ. Distinct pathways regulated by RET and estrogen receptor in luminal breast cancer demonstrate the biological basis for combination therapy. Ann Surg. 2014 Apr;259(4):793-9. doi: 10.1097/SLA.0b013e3182a6f552. PMID 24045439
- [Background] Spanheimer PM, Park JM, Askeland RW, Kulak MV, Woodfield GW, De Andrade JP, Cyr AR, Sugg SL, Thomas A, Weigel RJ. Inhibition of RET increases the efficacy of antiestrogen and is a novel treatment strategy for luminal breast cancer. Clin Cancer Res. 2014 Apr 15;20(8):2115-25. doi: 10.1158/1078-0432.CCR-13-2221. Epub 2014 Feb 13. PMID 24526731